CLINICAL TRIAL: NCT01771016
Title: Emergency Contraception - Observational Study of User's Profile
Brief Title: Emergency Contraception - User's Profile
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Principal Investigator, Kurt Hersberger, Prof., University Hospital, Basel, Switzerland
Other Study IDs: EKBB 114/07
Record Dates: First submitted 2013-01-14; First posted 2013-01-18 (Estimated); Last update posted 2013-01-18 (Estimated); Status verified 2013-01

CONDITIONS: Postcoital Contraception
Keywords: Emergency contraception; Emergency hormonal contraception; Community pharmacies; Pharmaceutical care; Time to access; Written assessments; Switzerland

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Retrospective analysis of requests of emergency hormonal contraception using pharmacy protocols registered in 2003 and 2006.

DETAILED DESCRIPTION:
In 2002, Levonorgestrel was introduced in Switzerland for emergency hormonal contraception (EC) without prescription ('pharmacist only'). In 2003, a first analysis of requests of EC showed that the dispensing of EC through pharmacies could successfully be implemented (Lemke et al 2004).

This study was repeated three years later with the aim to explore whether the user's profile has changed after introduction of a low threshold access to EC.

ELIGIBILITY:
Inclusion Criteria:

* women seaking emergency hormonal contraception

Exclusion Criteria:

-

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Pharmacies in Basle, Berne or Zurich, three major towns in the German speaking part of Switzerland, were purposively recruited if they had extended opening hours (emergency pharmacies) or if they were located downtown and open during traditional business hours (walk-in pharmacies).
  The pharmacists were asked if a pharmacy student could come to their place and photocopy the completed official one-page EHC written assessment forms.
Sampling Method: Non-Probability Sample
Enrollment: 729 (Actual)
Dates: Start 2006-01; Primary Completion 2008-12 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Sexual and protective behaviour | 2 years
  questions of interest: "Did you forget to take the pill?", "Did you have any other unprotected sexual intercourse since your last period?" and "Have you ever taken the "morning-after pill" before?"

SECONDARY OUTCOMES:
elapsed hours since unprotected intercourse | 1 month

OTHER OUTCOMES:
pharmacy status and care activity | 1 month
  pharmacy status (walk-in or emergency), and the three activities of the pharmacists (performance of a pregnancy test, delivery of EHC, referral to a physician).

CONTACTS AND LOCATIONS:
Overall Officials: Kurt E Hersberger, Prof., Principal Investigator — Dept Pharmaceutical Sciences, University Basel